CLINICAL TRIAL: NCT00169676
Title: Laparoscopic Radical Prostatectomy: A Registry and Database
Brief Title: Registry and Database Lap Prostatectomy
Status: Completed | Type: Observational
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: James Lingeman, MD, Methodist Urology
Other Study IDs: 03-040
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2008-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort: Registry and Database
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — registry and database for surgery outcomes

SUMMARY:
Recently, many centers have begun offering laparoscopic radical prostatectomy (LRP) as a minimally invasive therapy for localized prostate cancer.1-6 LRP may offer the advantages of improved neurovascular bundle sparing, a more precise urethrovesical anastomosis, shorter hospitalization, and decreased convalescence.

Our group at Methodist Urology, LLC has extensive experience in laparoscopy and in treating prostate cancer and are planning to offer LRP. We intend to maintain a registry and database to document the outcomes with LRP.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer death in men today. An estimated 220,900 new cases will be diagnosed in 2003 according to the American Cancer Society.7 Prostate cancer will account for one-third of the new cancer diagnoses in men in 2003. Prostate specific antigen (PSA), a sensitive screening method for prostate cancer, has helped diagnose prostate cancer at earlier stages. Stamey et al. found that the diagnosis of prostate cancer in patients with T1c disease (no abnormalities on digital rectal examination but elevated PSA) increased from10% in 1988 to 73% in 1996 and the increase in organ confined cancers increased from 40% to 75% over the same time period.8

Current surgical options for organ confined prostate cancer include open radical retropubic prostatectomy, open radical perineal prostatectomy, radioactive seed implantation, and radiation therapy. Open radical retropubic prostatectomy was pioneered in 1947 by Millin but what was slow to gain widespread acceptance secondary to associated morbidity.9-13 Refinement of the retropubic approach by Walsh has greatly improved outcomes, making it the most common surgical approach for radical prostatectomy.14, 15

As with other procedures, interest in the laparoscopic approach for radical prostatectomy developed in hopes of minimizing patient morbidity. In 1992, Schuessler et al performed the first LRP but the technical difficulties of the procedure at that time prohibited the widespread application of this technique.16 In 1998, Guillonneau et al introduced the Mountsouris technique in which a transperitoneal approach was used to perform the LRP.17, 18 Other groups have used this approach and even adapted this technique to perform extraperitoneal approaches to LRP.1, 2, 4, 5, 19, 20 Many centers are currently offering LRP as primary therapy for organ confined prostate cancer.

All curative surgical therapies for prostate cancer, whether performed in an open or laparoscopic manner, can result in impotence and/or incontinence. Incontinence can be treated with simple measures, such as muscle strengthening exercises, or if more bothersome, can be treated with surgical therapy. Impotence can be treated with medications or, if needed, surgery.

The relative risk of having positive surgical margins in patients undergoing open radical retropubic prostatectomy compared to laparoscopic radical prostatectomy is not known. Preliminary publications regarding laparoscopic radical prostatectomy report rates of positive surgical margins (13-25%) that are similar to open radical prostatectomy (11-46%).2, 5, 6, 19, 21-28 However, long-term follow-up is not available for patients undergoing laparoscopic radical prostatectomy, so the impact of positive margins on long-term survival is not known.

ELIGIBILITY:
Inclusion criteria:

* Patient of Methodist Urology in Indianapolis, IN
* Ability to give informed consent
* Biopsy proven diagnosis of prostate cancer without local extension or metastatic disease (Clinical T2 or less in the TNM classification)

Exclusion criteria:

* Major abdominal surgery precluding a safe laparoscopic approach
* Bleeding diathesis or anticoagulation
* Medical disease (such as cardiovascular or pulmonary diseases) precluding general anesthesia/laparoscopy
* Transplanted kidney in the pelvis
* Radiation therapy to pelvis
* Morbid obesity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Methodist Urology that are scheduled to undergo a laser procedure for prostate removal
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2003-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To create a registry and database for the treatment of localized prostate cancer with LRP. To record long term outcomes for patients undergoing Laparoscopic Radical Prostatectomy. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Larry Munch, MD, Principal Investigator — Methodist Urology, LLC
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States